CLINICAL TRIAL: NCT03877666
Title: Intraoperative Assessment of the Influence of Cleft Repair on Microcirculation of the Palate
Brief Title: Assessment of the Influence of Cleft Repair on Microcirculation of the Palate
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Microcirculation Palate
Record Dates: First submitted 2019-03-11; First posted 2019-03-18 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Cleft Palate; Cleft Lip and Palate
MeSH Terms: conditions — Cleft Palate; Cleft Lip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Investigators aim to evaluate the influence of cleft surgery on the tissue microcirculation of the palate with a non-invasive measurement.

ELIGIBILITY:
Inclusion Criteria:

* patients with orofacial clefts, who undergo routine cleft repair

Exclusion Criteria:

* missing datasets
* no signed consent for research.

Ages: 6 Months to 13 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Patients with orofacial clefts undergoing surgical repair of the deformity.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-08-04 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in tissue perfusion (regional tissue oxygen saturation (StO2%)) before and after surgery non-invasively measured | One measurement before surgery, one measurement immediately after surgery
  The difference and impact of our routine surgical technique on the tissue perfusion of the palate is measured non-invasively with a probe (regional StO2%). Localized measurement of the microvascular hemoglobin oxygen saturation.

SECONDARY OUTCOMES:
Status of wound healing | at 3 month and 6 month after surgery
  status of wound healing, fistula formation

CONTACTS AND LOCATIONS:
Overall Officials: Benito K Benitez, MD DDS MHBA, Principal Investigator — University Basel and University Hospital Basel
Locations (1):
- Universitätsspital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huang MH, Lee ST, Rajendran K. Clinical implications of the velopharyngeal blood supply: a fresh cadaveric study. Plast Reconstr Surg. 1998 Sep;102(3):655-67. doi: 10.1097/00006534-199809030-00007. PMID 9727428
- [Background] Mueller AA, Schumann D, Reddy RR, Schwenzer-Zimmerer K, Mueller-Gerbl M, Zeilhofer HF, Sailer HF, Reddy SG. Intraoperative vascular anatomy, arterial blood flow velocity, and microcirculation in unilateral and bilateral cleft lip repair. Plast Reconstr Surg. 2012 Nov;130(5):1120-1130. doi: 10.1097/PRS.0b013e318267d4fb. PMID 23096613
- [Background] Woo AS. Evidence-Based Medicine: Cleft Palate. Plast Reconstr Surg. 2017 Jan;139(1):191e-203e. doi: 10.1097/PRS.0000000000002854. PMID 28027255